CLINICAL TRIAL: NCT05046860
Title: Efficacy of Dalbavancin in Osteoarticular Infections Associated With Hip and Knee Replacements
Acronym: PRODALBA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-AOI-03
Record Dates: First submitted 2021-09-13; First posted 2021-09-16 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Osteoarticular Infection
Keywords: hip prosthese; knee prosthese
MeSH Terms: interventions — dalbavancin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dalbavancine + Rifampicine (Experimental)
  Interventions: Drug: Dalbavancin

INTERVENTIONS:
Drug: Dalbavancin — The unit dose of dalbavancin administered via the peripheral venous route will be 1500 mg at each injection with a first injection at Day1, a second injection at Day15 and a third at Day36, which corresponds to 61 days of treatment with dalbavancin.
  In case of residual dalbavancin dosage at Day15 lower than 15 mg/L (rare situation) and a minimal inhibitory concentration for dalbavancin of 0.125mg/L (less than 5% of the strains), an injection every 14 days will be necessary, i.e. Day1, Day15, Day29, Day43 and Day57, which corresponds to 71 days of dalbavancin treatment.
  Rifampicin should be given orally at a dose of 600 mg on an empty stomach in the morning for patients weighing less than 70 kg and 900 mg on an empty stomach in the morning for patients weighing more than 70 kg.

SUMMARY:
Osteoarticular infections associated with hip and knee prostheses require optimal surgical and medical management to maximize the rate of therapeutic success. Antibiotic therapy should be administered for a period of 12 weeks. Tolerance problems, difficulties in maintaining compliance over 12 weeks, bacterial multidrug resistance and sometimes intravenous administration are the main obstacles to appropriate antibiotic therapy and to limiting iatrogenicity. Dalbavancin is an antibiotic derived from teicoplanin (glycopeptide) with a long half-life, of punctual parenteral administration without a central line, active on staphylococci, and well tolerated. The data in the literature concerning its efficacy in Osteoarticular infections associated with hip and knee prostheses are limited and heterogeneous. Investigators would like to describe its efficacy in a homogeneous series of patients in terms of the type of infection, their surgical management and the methods of administration of the product in order to extend its use.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* First monomicrobial osteoarticular infection of knee or hip prosthesis with staphylococcus sensitive to dalbavancin (determined by a minimum inhibitory concentration by microdilution of the strain in question for vancomycin less than or equal to 2mg/L) and rifampicin, treated surgically by debridement, antibiotics and implant retention with change of moving parts (acute infections) or change in 1 stage (chronic infections)
* Social security affiliation
* Signature of informed consent

Exclusion Criteria:

* Hypersensitivity to glycopeptides or rifampin or to any of the excipients
* Porphyrias
* Probabilistic antibiotic treatment not administered within 24 hours of surgery
* Probabilistic antibiotic treatment that did not take into account the bacterium causing the infection in its spectrum
* Acute hematogenous infection (acute secondary)
* Use of background treatment incompatible with the inducing effect of rifampicin (see Summary of Product Characteristics for rifampicin)
* Contraindications to rifampin therapy: Moderate to severe impairment of liver function, patients with a history of hypersensitivity to other rifamycins, porphyria.

Hepatic cirrhosis

* Use of ototoxic therapy, such as an aminoglycoside
* Renal function with glomerular filtration rate less than 30 ml/min as measured by MDRD (Modification of Diet in Renal Disease)
* Pregnant and breastfeeding women: at inclusion a blood pregnancy test will be performed for women of childbearing age. The results will be communicated to the patient by a physician of her choice.
* Women of childbearing age not using an effective method of contraception (pill, intrauterine device, vaginal ring, contraceptive skin patch, hormonal subcutaneous implant, surgical sterilization)
* Protected persons defined in the following articles of the public health code:

L. 1121-6: persons deprived of liberty by a judicial or administrative decision, persons hospitalized without consent and persons admitted to a health or social establishment for purposes other than research; L. 1121-8: adults subject to a legal protection measure or unable to express their consent; L. 1122-1-2: persons in emergency situations who are unable to give prior consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
therapeutic success | 12 months
  therapeutic success defined by the absence of failure within 12 months of surgical management

SECONDARY OUTCOMES:
therapeutic success at 24 months | 24 months
  therapeutic success defined by the absence of failure within 24 months of surgical management
Tolerance | 6 months of first administration of dalbavancin
  Tolerance will be assessed by collecting adverse events during treatment with dalbavancin and rifampin classified according to Common Terminology Criteria for Adverse Events (version 5.0) within 6 months of its first administration.
Residual dalbavancin dosage | Day 61 of first administration of dalbavancin
  Residual dalbavancin dosage at Day61

CONTACTS AND LOCATIONS:
Overall Officials: Aurélien DINH, MD, Principal Investigator — AP-HP - Hôpital Ambroise-Paré; Eric SENNEVILLE, PD, Principal Investigator — Centre Hospitalier de Tourcoing
Locations (4):
- France (4):
  - AP-HP - Hôpital Ambroise-Paré, Boulogne-Billancourt
  - CHU de Nice, Nice
  - Centre Hospitalier de Tourcoing, Tourcoing
  - CHRU de TOURS, Tours